CLINICAL TRIAL: NCT04955197
Title: Accuracy of Exfoliated Cytology in Detection of Oral Premalignant and Malignant Lesions
Brief Title: Exfoliated Cytology in Detection of Oral Premalignant and Malignant Lesions
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mostafa Hassan Elnaggar, assistant lecturer, Cairo University
Other Study IDs: Cancer screening
Record Dates: First submitted 2021-07-04; First posted 2021-07-08 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Oral Cancer; Diagnoses Disease
Keywords: diagnosis; screening
MeSH Terms: conditions — Mouth Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the histo-pathological picture: In the present study, the exfoliated cytology of group II and III will be compared to the histo-pathological picture of the lesion "reference standard". That is because the histopathology analysis is the definitive diagnosis of oral mucosal lesions
  Interventions: Diagnostic Test: exfoliated cytology

INTERVENTIONS:
Diagnostic Test: exfoliated cytology — Micronuclei (MN) are small chromatin bodies in the cytoplasm formed by chromosome fragments or whole chromosomes that fail to be included in the nuclei during cell division. They are considered as a sensitive indicators of genetic damage. They are usually found in the basal cells of epidermis and are shed as exfoliated cells on maturation. Hence micronuclei assay can be used as monitoring of genetic damage, as it is increased in oral neoplastic conditions. Consequently, detection of micronuclei in exfoliated cells indicates an increased risk for cancer

SUMMARY:
Micronuclei have been used since 1937 as an indicator of genetic toxic exposure due to their association with chromosomal alterations. They can be detected in exfoliated cells and used as an indicator of recent DNA injury within oral mucosa. The buccal epithelial cells are first to be interacted with the cancer compounds such as tobacco (nicotine), which in turn induces the frequency of micronuclei under the influence of saliva. The exfoliated cell micronuclei assay involves microscopic analysis of oral smears to determine the prevalence of micro-nucleation. The assay is reliable and technically easy to perform, noninvasive and sensitive with limited cost.

DETAILED DESCRIPTION:
The study will be held at the Faculty of Dentistry Cairo University and the NCI All the participants will be administrated a standardized questionnaire to obtain demographic data, medical records and any history of relevant risk factors. The detailed clinical examination will be performed on each patient to assess the site, size, and the clinical characteristics of the lesion as well as the extent of local infiltration (if any) and cervical lymph node metastases (if any).

The entire procedure will be explained to the patients and an informed consent will be obtained. The participants were asked to rinse their mouth thoroughly with tap water 2-3 times immediately before the sampling procedure to reduce the oral bacterial load. Pre-moistened separate wooden spatula was used to scrape the oral buccal mucosa cells (right and left buccal mucosal cells). The cells were then smeared over clean, coded glass slides. The slides were then air dried and fixed in fixative for 20 minutes and stained. Afterwards the glass slide was rinsed with aqua dest and dried in the air. The slides will be prepared for microscopic analysis The criteria parameters for identifying micronucleus:

* Rounded smooth perimeter suggestive of a membrane.
* Less than one-third the diameter of the associated nucleus, but large enough to discern shape and color.
* Staining intensity similar to the nucleus.
* Texture similar to the nucleus.
* Same focal plane as the nucleus.
* Absence of overlap with or bridge to the nucleus.

Dead or degenerating cells (karyolysis, karyorrhexis, nuclear fragmentation) were excluded from the evaluation. Incisional or excisional biopsy will be obtained from subjects diagnosed with premalignant lesions and histo-pathological examination will be performed as an additional supportive test .

ELIGIBILITY:
Inclusion Criteria:

* Control group I: Participants with clinically normal oral mucosa and no evidence of any cancer risk factor as smoking and alcohol consumption.
* Control group II: Participants with clinically normal oral mucosa and with evidence of any cancer risk factor as smoking and alcohol consumption.
* Compare group III: Participants with potentially malignant lesions
* Compare group IV: Participants diagnosed with malignant disorders.
* All age range will be included irrespective of their sex.

Exclusion Criteria:

* • Individuals who had a recent viral infection or had undergone radiation therapy.

  * Those patients were excluded from the control group who had any history of tobacco intake or alcohol consumption and under medications.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants with clinically normal oral mucosa and no evidence of any cancer risk factor as smoking and alcohol consumption.Participants with clinically normal oral mucosa and with evidence of any cancer risk factor as smoking and alcohol consumption. Participants with potentially malignant (leukoplakia, oral lichen planus, smoker keratosis and erythroplakia) Participants diagnosed with malignant disorders.
  • All age range will be included irrespective of their sex.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Micronuclei presence | 5 minutes
  a sensitive indicators of genetic damage. They are usually found in the basal cells of epidermis and are shed as exfoliated cells on maturation. Hence micronuclei assay can be used as monitoring of genetic damage, as it is increased in oral neoplastic conditions.

CONTACTS AND LOCATIONS:
Overall Officials: alaa elnaggar, MSD, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jadhav K, Gupta N, Ahmed MB. Micronuclei: An essential biomarker in oral exfoliated cells for grading of oral squamous cell carcinoma. J Cytol. 2011 Jan;28(1):7-12. doi: 10.4103/0970-9371.76941. PMID 21552400